CLINICAL TRIAL: NCT06997926
Title: Identification of the Mechanism of Non-histaminergic Itch Probing Epigenetic Changes Following Cowhage Application
Brief Title: Identification of the Mechanism of Non-histaminergic Itch Inducing Epigenetic Changes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20220025
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Itch
MeSH Terms: conditions — Pruritus | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Two groups of subjects: one group will receive active cowhage spicules (itch inducer) and the other group will receive inactivated cowhage spicules (control)
Who Masked: Participant
Masking Description: The participants are blinded about receiving active or inactive cowhage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cowhage (Active Comparator): The participant will receive active cowhage in the forearm.
  Interventions: Procedure: blood sampling
- Inactive cowhage (Sham Comparator): The participant will receive inactive cowhage in the forearm.
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — Whole blood samples (5 mL per each time point, a total of 20 mL per subject) will be collected

SUMMARY:
Itch is defined as an unpleasant sensation that evokes the desire to scratch. Chronic itch, defined as itch persisting for more that 6 weeks, is a key symptom in many diseases severely affects the quality of life of the affected patients and represents a substantial economic burden for the society. At present, there are no effective treatments for chronic itch diseases. Moreover, chronic itch patients express differences in their genes compared with people who do not suffer from itch.

With this experiment, we wish to analyse differences in genes expression in healthy volunteers who have been exposed to artificial itch from small plant needles from the plant cowhage (mucuna pruriens) and compare them to controls who have not been exposed to itch.

DETAILED DESCRIPTION:
The study takes place over 2 sessions over a period of 2 days. Thirty healthy participants will be randomly allocated into two groups named "active group", treated with active cowhage spicules, and "control group", exposed to inactivated cowhage spicules.

During the 1st session, the participant will fill out a questionnaire including basic information and after participants in the active group will be treated with cowhage spicules for 15 minutes, while participants in the control group will receive the inactivated cowhage spicules. All subjects will be provided with a visual analog scale in which they have to report continuously the sensation of itch and pain on a scale from 0 to 100 for 15 minutes. Before cowhage application, 30 minutes and 3 hours after cowhage application, blood samples will be collected from all participants. The 2nd session will take place 24 h after the 1st session and in this session the final blood sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* 18-60 years
* Speak and understand English

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction defined as any use of cannabis, opioids, or other addictive drugs
* Previous or current history of neurological (e.g., neuropathy), immunological (e.g., asthma, immune deficiencies, arthritis) musculoskeletal (e.g., muscular pain in the upper extremities), cardiac disorder, or mental illnesses that may affect the results,
* Lack of ability to cooperate
* Current use of medications that may affect the trial such as antihistamines, antipsychotics, and pain killers, as well as systemic or topical steroids

  * Allergy to lidocaine
  * Skin diseases (e.g., atopic dermatitis, pruritus nodularis, eczema, psoriasis)
  * Moles, scars, or tattoos in the area to be treated or tested.
  * Consumption of alcohol or painkillers 24 hours before the study days and between these
  * Smoking
  * Acute or chronic pain
  * Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
miRNA expression over time | Before active/inactive cowhage
  Plasma miRNA evaluation
miRNA expression over time | 30 minutes post-Active/inactive cowhage
  Plasma miRNA evaluation
miRNA expression over time | 3 hours post-active/inactive cowhage
  Plasma miRNA evaluation
miRNA expression over time | 24 hours post-active/inactive cowhage
  Plasma miRNA evaluation
Protein expression over time | Before active/inactive cowhage
  Plasma protein evaluation
Protein expression over time | 30 minutes post-active/inactive cowhage
  Plasma protein evaluation
Protein expression over time | 3 hours post-active/inactive cowhage
  Plasma protein evaluation
Protein expression over time | 24 hours post-active/inactive cowhage
  Plasma protein evaluation

SECONDARY OUTCOMES:
Assessment of itch: visual analog scale (VAS) | Immediately after Active/inactive cowhage
  Itch following pruritogens will be monitored for 15 minutes using a computerized 100 mm visual analog scale (eVAS software Aalborg University, Denmark), installed on a tablet. The scale range from 0 (no itch) to 100 (worst imaginable itch).
Assessment of pain: visual analog scale (VAS) | Immediately after Active/inactive cowhage
  Pain following pruritogen will be monitored for 15 minutes using a computerized 100 mm visual analog scale (eVAS software Aalborg University, Denmark), installed on a tablet. The scale range from 0 (no pain) to 100 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Gistrup, Denmark

IPD SHARING:
Plan to Share IPD: No